CLINICAL TRIAL: NCT02561182
Title: Bone Health in Patients With Overgrowth
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Megha M. Tollefson, M.D., PI, Mayo Clinic
Other Study IDs: 15-002284
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Bone Mineral Density; Vascular Malformations
MeSH Terms: conditions — Vascular Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients aged 5 years old and with a known diagnosis of a OGS

SUMMARY:
The goal of this study is to determine whether or not patients with overgrowth syndromes have decreased bone density.

DETAILED DESCRIPTION:
It is known that patients with complex vascular malformation are at risk of decreased bone density and even vanishing bone disease. However, what is not known is if patients with OGS are at decreased bone density at locations that are distant from the vascular malformation.

This study will look at bone health in patient's with OGS in a cross sectional fashion. If they are found to be at a particular risk for decreased bone density then this can be addressed in early childhood, through nutrition and activity recommendations.

The study will consist of 15 participants, all who have a known clinical diagnosis of an overgrowth syndrome, and will be >5 years old so that they can co operate with a DEXA or Xtreme CT scan.

Study specifics:

* They will be asked specific questions regarding medical and family history and an intake form will be filled out.
* The height, weight, body mass index and Tanner stage measurements will be recorded during this visit.
* Photos of the affected area(s) will be taken, however, this is optional.
* A urine pregnancy test will be done in all females of childbearing potential .
* Laboratory studies will be performed in all patients.
* A 24-hour urine sample will be collected from adults who are able and willing; in children and in those not able or unwilling to provide a 24-hour urine, a spot urine will be collected.
* Bone age will be assessed via plain film of the wrist
* Bone density will be assessed for each patient via DEXA scan
* Cortical and trabecular parameters and bone strength will be assessed by HRpQCT

ELIGIBILITY:
Inclusion Criteria:

* Age > 5 years such that the patient is able to cooperate with the DXA scan or Xtreme CT
* Known clinical diagnosis of an overgrowth syndrome such as Klippel-Trenaunay Syndrome, CLOVE syndrome, Proteus syndrome, diffuse capillary malformation with overgrowth, or other unspecified OGS.

Exclusion Criteria:

* Age < 5 years
* Inability to comply with the scan
* No or uncertain diagnosis of an OGS.
* Prior bisphosphonate use
* Systemic steroids in the past 6 months
* Pregnant women

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 5 years old and over with a known clinical diagnosis of an overgrowth syndrome such as Klippel-Trenaunay Syndrome, CLOVE syndrome, Proteus syndrome, diffuse capillary malformation with overgrowth, or other unspecified OGS.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-09; Primary Completion 2019-05-23 (Actual); Study Completion 2019-05-23 (Actual)

PRIMARY OUTCOMES:
Evidence of decreased bone density in patients with vascular malformations, confirmed by DEXA scans | One year
Evidence of decreased bone density in patients with vascular malformations, confirmed by serum specific bone markers | One year
  Bone markers : Alkaline phosphatase; albumin; PTH; 1-25 dihydroxyvitamin D, 25- hydroxyvitamin D

CONTACTS AND LOCATIONS:
Overall Officials: Megha M Tollefson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials